CLINICAL TRIAL: NCT04985617
Title: The Effects of Active Warming on Temperature on Core Body and Thermal Comfort in Patients After Transurethral Resection of The Prostate
Brief Title: The Effects of Active Warming on Temperature on Core Body and Thermal Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, HÜLYA YILMAZ, PhD, Principal Investigator, Msc, PhD Hülya YILMAZ, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08/02/2019- E.43649
Record Dates: First submitted 2021-07-16; First posted 2021-08-02 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Hypothermia; Thermal Comfort; Body Temperature Changes
Keywords: fluid infusion; postoperative hypothermia; nursing; active warming
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized controlled experimental study.
Masking Description: The intervention and measurements were carried out by the first researcher, and the patients discovered their own groups when the postoperative warming intervention was applied to them. Because of the nature of the intervention, blinding could not be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warmed Fluids (Experimental): When patients recovered from the effect of anesthesia, awakened and were able to switch to normal spontaneous breathing, they were taken from the sober unit to the service or intensive care unit, and subsequent follow-ups were carried out by the researcher in these units. The IV fluid given to the patients in the intervention group was heated to 36ºC using the medical heating device.
  Interventions: Other: Warmed Fluids
- Room Temperature Fluids (No Intervention): When patients recovered from the effect of anesthesia, awakened and were able to switch to normal spontaneous breathing, they were taken from the sober unit to the service or intensive care unit, and subsequent follow-ups were carried out by the researcher in these units. The IV fluid given to the patients in the control group was given at room temperature without heating and without intervention

INTERVENTIONS:
Other: Warmed Fluids — The IV fluid given to the patients in the intervention group was heated to 36ºC using the medical heating device.
  Arms: Warmed Fluids

SUMMARY:
Purpose: This study was conducted to examine the effect of warmed intravenous fluids (WIVF) on the core body temperature and the patients' thermal comforts during the postoperative period in patients undergoing transurethral resection of the prostate (TURP).

Design: This was a prospective, randomized controlled experimental study. Methods: A total of 105 male patients undergoing TURP surgery and bladder irrigation were randomized to one of either room temperature (n=51) or warmed intravenous fluids (n=54) groups in postanesthesia care unit. The fluids in the experimental group were warmed until the body temperature was reached 36.0°C.

DETAILED DESCRIPTION:
Purpose: This study was conducted to examine the effect of warmed intravenous fluids (WIVF) on the core body temperature and the patients' thermal comforts during the postoperative period in patients undergoing transurethral resection of the prostate (TURP).

Design: This was a prospective, randomized controlled experimental study. Methods: A total of 105 male patients undergoing TURP surgery and bladder irrigation were randomized to one of either room temperature (n=51) or warmed intravenous fluids (n=54) groups in postanesthesia care unit. The fluids in the experimental group were warmed until the body temperature was reached 36.0°C. The intravenous (IV) fluid given to the two groups was 1000 ml of 0.9% isotonic sodium chloride solution.

ELIGIBILITY:
Inclusion Criteria:

* patients who age bigger than18,
* patients who were undergoing general anesthesia, to whom voluntary hypothermia was not applied during the operation,
* patients who were hemodynamically stable,
* patients who had a physician's order for 1000 ml of 0.9% Isotonic Sodium Chloride IV fluid treatment,
* patients were undergoing bladder irrigation were included in the study.
* patients the sense, expression of heat by the patient in recovery,
* patient who accepted to participate to the study

Exclusion Criteria:

* patients have any infection, fever
* patients have underlying diseases (hypothyroidism, hyperthyroidism, diabetes, cardiovascular disease or kidney failure)
* patients who had mental deficiency that could prevent communication,
* patients who had visual or hearing impairments,
* patients who were receiving mechanical ventilation support, were sedated,
* patients were the need for open surgery or any reason for returning the patient to the operating room,
* patients need for postoperative blood transfusions,
* patients have intra-abdominal infection,
* patients have an unexpected allergy to anesthetic drugs,
* patients have a temperature higher than 36.0ºC,
* patients have for cardiopulmonary resuscitation,
* patients have severe hemodynamic changes during the operation.

Ages: 37 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Bening prostatic hyperplasia (BPH) is a histopathological condition requiring surgical intervention in men over 60 years of age due to the increase or proliferation of epithelial and stromal tissues of the prostate around the urethra (Dirim, 2010; Gilroy, 2015).
Enrollment: 105 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Thermal Comfort Scale (TCS) | 6 months
  Thermal Comfort Scale (TCS): This is a Likert type scale which was developed by Wagner et. al. (2006) and the validity and reliability in Turkish was tested by Özsaban (2017). The evaluation of thermal comfort was made by the face to face interview method for all patients. The TCS evaluates the patient's temperature comfort perception subjectively. The scale consists of 13 items in total, and each item is scored between 1 and 6 points. A high score indicates a high temperature comfort level.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Health Sciences Institute, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When patients recovered from the effect of anesthesia, awakened and were able to switch to normal spontaneous breathing, they were taken from the sober unit to the service or intensive care unit, and subsequent follow-ups were carried out by the researcher in these units. The IV fluid given to the patients in the intervention group was heated to 36ºC using the medical heating device, and the IV fluid given to the patients in the control group was given at room temperature without heating. The environment temperature of the room was the same in the service, intensive care, and recovery units on the same day. The environment temperature of the room varied between 20ºC and 25ºC on the different days on which the research was implemented. The air humidity level was between 32% and 45%. Body temperature was measured as soon as the infusion started and was repeated every 60 minutes using a "tympanic thermometer".
Supporting Information: Study Protocol
Time Frame: 6months
Access Criteria: Active Warming on Temperature on Core Body and Thermal Comfort in Patients

REFERENCES:
- [Background] Xu HX, You ZJ, Zhang H, Li Z. Prevention of hypothermia by infusion of warm fluid during abdominal surgery. J Perianesth Nurs. 2010 Dec;25(6):366-70. doi: 10.1016/j.jopan.2010.10.007. PMID 21126666
- [Background] Woolnough M, Allam J, Hemingway C, Cox M, Yentis SM. Intra-operative fluid warming in elective caesarean section: a blinded randomised controlled trial. Int J Obstet Anesth. 2009 Oct;18(4):346-51. doi: 10.1016/j.ijoa.2009.02.009. Epub 2009 Aug 7. PMID 19665366
- [Background] Chung SH, Lee BS, Yang HJ, Kweon KS, Kim HH, Song J, Shin DW. Effect of preoperative warming during cesarean section under spinal anesthesia. Korean J Anesthesiol. 2012 May;62(5):454-60. doi: 10.4097/kjae.2012.62.5.454. Epub 2012 May 24. PMID 22679543
- See also: Prevention of hypothermia by infusion of warm fluid during abdominal surgery — https://doi.org/10.1016/j.jopan.2010.10.007
- See also: Intra-operative fluid warming in elective caesarean section: a blinded randomised controlled trial — http://doi.org/10.1016/j.ijoa.2009.02.009
- See also: Effect of preoperative warming during cesarean section under spinal anesthesia. — http://doi.org/10.4097/kjae.2012.62.5.454